CLINICAL TRIAL: NCT06855147
Title: A Single-center, Open-label, Phase Ⅰ Clinical Study of the Absorption, Metabolism, and Excretion of [14C]HRS9531 in Healthy Male Subjects
Brief Title: Mass Balance Study of [14C]HRS9531 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-109
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]HRS9531 Group (Experimental)
  Interventions: Drug: [14C]HRS9531

INTERVENTIONS:
Drug: [14C]HRS9531 — A single dose of [14C]HRS9531 injected subcutaneously.

SUMMARY:
This study was a single-center, single-dose, open-label study in healthy male subjects to investigate the absorption, metabolism and excretion of HRS9531 after a single subcutaneous injection of [14C]HRS9531.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form prior to the trial and have a full understanding of the trial's procedures, content and potential adverse reactions.
2. Healthy male subjects aged between 18 and 55 years (inclusive), determined at the time of signing the informed consent.
3. Body weight ≥50 kg, and the body mass index (BMI) between 19 to 32.5 kg/m2.
4. From the signing of the informed consent form until 12 months after the last administration, the subject (including partner) has no family planning and is willing to use the high-efficiency contraceptive measures specified in the plan.

Exclusion Criteria:

1. History of any clinically important disease or disorder.
2. History of drug or other allergies, or who, in the judgement of the investigator, may be allergic to the study drug or any component of the study drug.
3. Physical examination, vital signs or other laboratory measurements, other electrocardiographic parameters, abdominal ultrasound (except mild fatty liver), and abnormalities on chest radiography as judged by the investigator to be clinically significant.
4. The subject was considered by the investigator to have any other factors that would preclude him from participating in the study or the subject withdrew from the study due to his own reasons.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax). | 0 to anticipated 64 days.
Time to reach the maximum concentration (Tmax). | 0 to anticipated 64 days.
Half-life (t1/2). | 0 to anticipated 64 days.
Total radioactive recovery rate in urine. | 0 to anticipated 64 days.
Total radioactive recovery rate in feces. | 0 to anticipated 64 days.
Cumulative radioactive recovery rate in urine. | 0 to anticipated 64 days.
Cumulative radioactive recovery rate in feces. | 0 to anticipated 64 days.

SECONDARY OUTCOMES:
Whole blood total radioactivity (TRA) ratio. | 0 to anticipated 64 days.
Plasma total radioactivity (TRA) ratio. | 0 to anticipated 64 days.
Adverse events (AEs). | 0 to 7 days after the last sample collection.
Serious adverse events (SAEs). | 0 to 7 days after the last sample collection.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided